CLINICAL TRIAL: NCT06746779
Title: Hisar Hospital Intercontinental
Brief Title: The Role of Preoperative Ureteral Diameter Measurements in Predicting Difficult Access During Retrograde Intrarenal Surgery: A Retrospective Analysis of 234 Patients
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Principal Investigator, Hisar Intercontinental Hospital
Other Study IDs: 13.12.2024. 24-12
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Kidney Stones; Retrograde Intrarenal Surgery; Difficult Ureteral Access Prediction
Keywords: Retrospective analysis of 234 patients undergoing retrograde intrarenal surgery (RIRS).
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easy Access Group: Patients with successful ureteral access on the first attempt during retrograde intrarenal surgery (RIRS).
- Difficult Access Group: Patients requiring multiple attempts for ureteral access, alternative procedures, or cases where the planned surgery could not be completed due to access issues.

SUMMARY:
This study investigates the role of preoperative ureteral diameter measurements in predicting difficult access during retrograde intrarenal surgery (RIRS) in patients with kidney stones. A retrospective analysis was conducted on 234 patients who underwent RIRS, evaluating factors such as preoperative ureteral diameters (measured at distal, iliac, and upper ureteral levels via CT scans), stone size, patient demographics, operation duration, and surgical success rates. The findings aim to determine whether ureteral diameter measurements can serve as reliable predictors for surgical challenges, ultimately improving preoperative planning and patient outcomes.

DETAILED DESCRIPTION:
This retrospective study evaluates the role of preoperative ureteral diameter measurements in predicting difficult access during retrograde intrarenal surgery (RIRS) in patients with kidney stones. A total of 234 patients who underwent RIRS were included in the analysis. Preoperative computed tomography (CT) scans were used to measure ureteral diameters at three levels: distal ureter, iliac ureter, and upper ureter. The relationship between ureteral diameter and intraoperative access difficulty was assessed.

The study also analyzed patient demographics (age, gender, BMI), stone characteristics (size, location), operative parameters (duration, access attempts), and outcomes (surgical success and complication rates). Difficult access during RIRS was defined based on the number of attempts required to achieve successful ureteral access, need for secondary procedures, or inability to complete the planned surgery.

The primary aim was to determine whether preoperative ureteral diameter measurements can serve as predictive markers for challenging surgical access. Secondary objectives included identifying other patient or stone-related factors contributing to access difficulty and evaluating their impact on surgical outcomes. The findings may assist clinicians in preoperative planning, improving patient selection for RIRS, and optimizing intraoperative strategies to minimize complications and enhance procedural success rates.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older. Diagnosed with kidney stones (nephrolithiasis) requiring surgical intervention. Underwent retrograde intrarenal surgery (RIRS). Available preoperative CT scans for ureteral diameter measurements. Complete medical records, including demographic, clinical, and surgical data.

Exclusion Criteria:

History of open or laparoscopic renal surgery. Presence of ureteral strictures or congenital anomalies. Patients with incomplete or missing medical records. Active urinary tract infection at the time of surgery. Pregnant or lactating individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years and older) who underwent retrograde intrarenal surgery (RIRS) for the management of kidney stones at a tertiary care center. Patients included in the study were evaluated retrospectively, with data obtained from their medical records, including preoperative imaging, intraoperative findings, and postoperative outcomes.
  The population represents a diverse group in terms of age, gender, body mass index (BMI), and stone characteristics (e.g., size, location). Patients with sufficient preoperative imaging data and complete surgical records were included to ensure accurate analysis of ureteral diameter measurements and their relationship to surgical outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Predictive Value of Preoperative Ureteral Diameter for Difficult Access During RIRS | Intraoperative (assessed during the surgical procedure).
  Evaluate the correlation between preoperative ureteral diameters (measured at distal, iliac, and upper ureteral levels via CT imaging) and the difficulty of achieving ureteral access during retrograde intrarenal surgery (RIRS).

CONTACTS AND LOCATIONS:
Overall Officials: Basri Cakiroglu, Principal Investigator — Hisar Intercontinental Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Basri Cakiroglu, Istanbul
  - Hisar Intercontinental Hospital, Istanbul